CLINICAL TRIAL: NCT07209735
Title: Effectiveness of the MINUTES Bundle for Initial 30-Minute Management of Undifferentiated Circulatory Shock in the Emergency Department
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omnia Esaam Abdelhady, Effectiveness of the MINUTES Bundle for Initial 30-Minute Management of Undifferentiated Circulatory Shock in the Emergency Department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MINUTES-SHOCK-2025
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Validation of Minute Bundle in Undifferntiated Shock
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to one of two parallel groups. The intervention group will receive the MINUTES bundle for the initial 30-minute management of undifferentiated circulatory shock in the emergency department, while the control group will receive standard care according to current departmental protocols. Outcomes will be compared between both groups to evaluate the effectiveness of the MINUTES bundle.
Masking Description: This is an open-label trial. Due to the nature of the intervention (implementation of the MINUTES bundle in the emergency department), blinding of participants, care providers, and investigators is not feasible.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants will receive the Minute Bundle, a structured package of early resuscitation interventio (Experimental)
  Interventions: Device: Ultrasound
- Participants will receive standard resuscitation according to current institutional protocols and tr (Active Comparator)
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Participants in this arm will receive the structured MINUTES bundle during the first 30 minutes of shock management in the emergency department. The bundle includes: continuous monitoring, intravenous access and fluid resuscitation, early initiation of norepinephrine when indicated, point-of-care ultrasound assessment (cardiac, IVC, and lung ultrasound) to guide diagnosis and resuscitation, essential laboratory tests, early antibiotics if infection is suspected, and source control or stabilization measures.

SUMMARY:
This study aims to validate the effectiveness of the MINUTES bundle on clinical outcomes in patients presenting with undifferentiated shock.

DETAILED DESCRIPTION:
Undifferentiated circulatory shock represents a critical challenge in emergency medicine (1), requiring rapid assessment and immediate intervention to prevent organ failure and death. Early goal-directed therapy (EGDT) and time-sensitive bundles have proven beneficial in improving outcomes. While specific shock types (e.g., septic, cardiogenic) have established guidelines (2-6), there is limited structured guidance for the initial 30-minute management "golden half hour" of resuscitation when the cause is unknown.

The MINUTES bundle, proposed in recent expert opinion (7), offers a structured approach to streamline early resuscitation and evaluation steps. It includes:

* Maintain ABCs (airway, breathing, circulation)
* INfuse vasopressors/fluids and INvestigate basic labs
* Ultrasound (POCUS)
* Treat underlying Etiology
* Stabilize systemic perfusion

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults 18-65 years old

  2. Clinical signs of circulatory shock:
  * SBP <90 mmHg or MAP <65 mmHg
  * Signs of hypoperfusion (altered mental status, oliguria, elevated lactate) 3. No clear etiology of shock at time of triage

Exclusion Criteria:

* 1- Trauma-related shock 2- Known terminal illness- Transferred after prior resuscitation 4- Pregnant patients 5-Patients with cardiac arrest upon arrival

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10-20 (Estimated)

PRIMARY OUTCOMES:
Shock reversal within 6 hours (MAP ≥65 mmHg without vasopressors + improved perfusion) | Minute bundle in initial 30-minute management Shock reversal within 6 hours